CLINICAL TRIAL: NCT00565799
Title: A Pilot Study of Metabolic Effects of Omentectomy in Obese Patients With Type 2 Diabetes Mellitus Treated With Laparoscopic Adjustable Gastric Banding (LAGB)
Brief Title: A Pilot Study of Metabolic Effects of Omentectomy
Acronym: OMT
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Conflicting interim data
Sponsor: NYU Langone Health (Other)
Collaborators: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 07-178
Record Dates: First submitted 2007-11-28; First posted 2007-11-30 (Estimated); Last update posted 2015-11-20 (Estimated); Status verified 2015-11

CONDITIONS: Patients Who Consented to Undergo Laparoscopic Gastric Banding Surgery for Weight Loss and Consent to Participate in This studyBMI ≥35 kg/m2; Confirmed Type 2 Diabetes Treated With Oral Agents and/or Only Diet Therapy; Age 18-64 Years
Keywords: DM

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1. Omentectomy (Active Comparator): LAGB & Omentectomy
  Interventions: Procedure: Omentectomy
- 2 No Omentectomy (Placebo Comparator): LAGB Only
  Interventions: Other: No intervention

INTERVENTIONS:
Procedure: Omentectomy — Removing the omentum
  Arms: 1. Omentectomy
Other: No intervention — Only LAGB without Omentectomy
  Arms: 2 No Omentectomy

SUMMARY:
PROTOCOL SUMMARY

Type of Study: Pilot, randomized and single center trial Test Procedure: Omentectomy Aim 1. Determine the effect of omentectomy on 1) insulin sensitivity, 2) beta cell function and 3) plasma markers of inflammation We hypothesize that removal of omental fat increases insulin sensitivity and pancreatic sensitivity to glucose, and decreases systemic inflammation.

Aim 2. Identify genes and proteins in adipocytes from obese patients that affect clinical presentation versus those that are affected by obesity for future study.

We hypothesize that the genetic samples will help us to identify genes and proteins in adipocytes from obese patients that affect clinical presentation versus those that are affected by obesity and help us to design future obesity genetic studies.

Total Enrollment Number: 30 patients who are scheduled to undergo bariatric surgery for weight loss at New York University Medical Center will be invited to participate in this study. Subjects will be randomly assigned, by using a computer-generated randomization scheme, in a single-blind fashion to either the omentectomy (n=15) or control group (n=15).

DETAILED DESCRIPTION:
Inclusion Criteria:

* Patients who consented to undergo LAGB for weight loss and consent to participate in this study
* BMI ≥35 kg/m2
* Confirmed T2DM treated with oral agents and/or only diet therapy
* Age 18-64 years

Exclusion Criteria:

* Insulin therapy
* Weight change (>2% body weight) within 4 weeks before surgery
* Patients with T2DM for more than 10 years

Research Design- Pilot Study Event Week (approximate) Medical Screening (in conjunction with routine pre-op visit) -4 OGTT & randomization -2 Preliminary genetic testing for the future study (blood sample) -2 Surgery with or without omentectomy 0 Preliminary genetic testing for the future study (fat sample) 0 Weight stabilization visit (in conjunction with routine post-op visit) 2 Weight stabilization visit (in conjunction with routine post-op visit) 4 OGTT 6

STUDY PLAN

Study has approved by IRB, NYU School of Medicine Committee, GCRC, and Bellevue Hospital.

Study initiation date: November 01, 2007

Enrollment period: Nov. 2007 to Nov. 2008

Study period: Nov. 2007 to Jan 2008

ELIGIBILITY:
Inclusion Criteria:

* Patients who consented to undergo LAGB for weight loss and consent to participate in this study
* BMI ≥35 kg/m2
* Confirmed T2DM treated with oral agents and/or only diet therapy
* Age 18-64 years

Exclusion Criteria:

* Insulin therapy
* Weight change (>2% body weight) within 4 weeks before surgery
* Patients with T2DM for more than 10 years

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2007-11; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
1) insulin sensitivity, 2) beta cell function and 3) plasma markers of inflammation | 6 week post op

SECONDARY OUTCOMES:
Identify genes and proteins in adipocytes from obese patients that affect clinical presentation versus those that are affected by obesity for future study. | 6 week post op

CONTACTS AND LOCATIONS:
Overall Officials: Christine Ren, M.D., Principal Investigator — NYU School of Medicine
Locations (1):
- NYU School of Medicine, New York, New York, United States

REFERENCES:
- See also: Related Info — http://nyuweightloss.org